CLINICAL TRIAL: NCT05797753
Title: A Phase 1, Single-center, Open-label, 2-part, 2-treatment Period, 1-sequence, Cross-over, Drug-drug Interaction Study to Investigate the Effect of Erythromycin on SAR443820 (Part A) and the Effect of Itraconazole on SAR443820 (Part B) in Healthy Adult Participants
Brief Title: A Study to Assess the Effect of Erythromycin on the Test Medicine (SAR443820) When Given Orally as Tablets to Healthy Adult Male and Female Participants (Part A); and the Effect of Itraconazole on the Test Medicine (SAR443820) When Given Orally as Capsules to Healthy Adult Male Participants (Part B)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INT17470; U1111-1267-9023 (Registry Identifier: ICTRP); INT17470 (Other: Sanofi Identifier)
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis; Healthy Volunteer
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Erythromycin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part-A, Period-1 (Experimental): Single dose of SAR443820 tablet on Day 1
  Interventions: Drug: SAR443820
- Part-A, Period-2 (Experimental): Single dose of SAR443820 tablet on Day 6, and erythromycin ethyl succinate (EES) three-time a day (TID) from Day 1 to Day 9
  Interventions: Drug: SAR443820; Drug: Erythromycin ethyl succinate
- Part-B, Period-1 (Experimental): Single dose of SAR443820 capsule on Day 1
  Interventions: Drug: SAR443820
- Part-B, Period-2 (Experimental): Single dose of SAR443820 capsule on Day 6, and Itraconazole once daily (QD) from Day 1 to Day 11
  Interventions: Drug: SAR443820; Drug: Itraconazole

INTERVENTIONS:
Drug: SAR443820 — Tablet by oral administration
  Arms: Part-A, Period-1; Part-A, Period-2
Drug: SAR443820 — Capsule by oral administration
  Arms: Part-B, Period-1; Part-B, Period-2
Drug: Erythromycin ethyl succinate — Tablet by oral administration
  Arms: Part-A, Period-2
Drug: Itraconazole — Capsule by oral administration
  Arms: Part-B, Period-2

SUMMARY:
This is a Phase 1, cross-over, 2-part study for pharmacokinetic (PK) assessment of SAR443820 when co-administered with cytochrome P450 3A4 (CYP3A4) inhibitors (erythromycin ethyl succinate (EES) in Part A and possibly itraconazole in Part B).

In Part A, the objective is to assess the effects of repeated administration of EES as CYP3A4 inhibitor, on the PK profile of a single oral dose of SAR443820 tablet in healthy male and female participants.

In Part B, the objective is to assess the effects of repeated administration of itraconazole on the PK profile of a single oral dose of SAR443820 capsule in healthy male participants.

Part A includes a screening period, Period 1 (SAR443820), a wash-out period and Period 2 (SAR443820 + EES). Part B includes a screening period, Period 1 (SAR443820), a wash-out period and Period 2 (SAR443820 + itraconazole). The washout period between single SAR443820 administration in Period 1 and the start of dosing with EES (Part A) or itraconazole (Part B) in Period 2 is at least 4 days.

The study duration is approximately 7 weeks for each Part A and Part B.

The treatment duration is:

* For SAR443820 (both Part A and Part B): 1 day in each Period; single dose of SAR443830 on Period 1 (P1)-Day 1 and on Period 2 (P2)-Day 6 for each Part.
* For EES (Part A): 9 days of treatment in Period 2 with P2-Day 1 starting at least 4 days after P1-Day 1.
* For itraconazole (Part B): the treatment duration lasts 11 days in Period 2 and it is fixed once the results of Part A are issued, P2-Day 1 starting at least 4 days after P1-Day 1.

DETAILED DESCRIPTION:
The study duration was approximately 7 weeks for each Part A and Part B.

ELIGIBILITY:
Inclusion Criteria:

* Part A: male or female participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent
* Part B: male participant only must be 18 to 55 years of age inclusive, at the time of signing the informed consent
* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index between 18.0 and 30.0 kg/m^2, inclusive
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), or infectious disease, or signs of acute illness - Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of hormonal contraception or menopausal hormone replacement therapy; any non-live Covid-19 vaccine within the last 2 weeks before inclusion, any live attenuated vaccine within the last 28 days before inclusion and any other non-vaccine biological drugs given within 4 months before inclusion
* Current enrollment in Part A (applicable for Part B) or past participation in previous clinical study on SAR443820
* Positive result for hepatitis B, C or human immunodeficiency virus (HIV)
* Positive result on urine drug screen
* Positive urine alcohol test
* Any consumption of citrus fruits (grapefruit, orange, etc) or their juices within 5 days before inclusion The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Part A: SAR443820: Area under the plasma concentration from time zero to the last concentration above the limit of quantification (AUClast) | Period 1: Day 1 to Day 3; Period 2: Day 6 to Day 10
Part A: SAR443820: Area under the plasma concentration (AUC) | Period 1: Day 1 to Day 3; Period 2: Day 6 to Day 10
Part B: SAR443820: AUClast | Period 1: Day 1 to Day 3; Period 2: Day 6 to Day 12
Part B: SAR443820: AUC | Period 1: Day 1 to Day 3; Period 2: Day 6 to Day 12

SECONDARY OUTCOMES:
Part A: SAR443820: Maximum plasma concentration observed (Cmax) | Period 1: Day 1 to Day 3; Period 2: Day 6 to Day 10
Part A: SAR443820: Time to reach Cmax (tmax) | Period 1: Day 1 to Day 3; Period 2: Day 6 to Day 10
Part A: SAR443820: Terminal half-life (t1/2z) | Period 1: Day 1 to Day 3; Period 2: Day 6 to Day 10
Part B: SAR443820: Cmax | Period 1: Day 1 to Day 3; Period 2: Day 6 to Day 12
Part B: SAR443820: tmax | Period 1: Day 1 to Day 3; Period 2: Day 6 to Day 12
Part B: SAR443820: t1/2z | Period 1: Day 1 to Day 3; Period 2: Day 6 to Day 12
Part A: Erythromycin ethyl succinate concentrations | Period 2: Day 6 and Day 7
Part A: Erythromycin base concentration | Period 2: Day 6 and Day 7
Part B: Itraconazole: Cmax | Period 2: Day 6 and Day 7
Part B: Itraconazole: AUClast | Period 2: Day 6 and Day 7
Part B: Hydroxyitraconazole: Cmax | Period 2: Day 6 and Day 7
Part B: Hydroxyitraconazole: AUClast | Period 2: Day 6 and Day 7
Part A: number of participants with treatment emergent adverse events (TEAEs) | Period 1: Day 1 to Day 4; Period 2: Day 1 to Day 10 + 3 days of end of study (EOS) period
Part B: number of participants with TEAEs | Period 1: Day 1 to Day 4; Period 2: Day 1 to Day 12 + 8-10 days of end of study (EOS) period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Nucleus Network Site Number : 8400001, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: INT17470 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25273&tenant=MT_SNY_9011